CLINICAL TRIAL: NCT06559969
Title: Randomized Controlled Study Comparing the Administration of Opioids Epidurally vs IV in Patients Undergoing Laparotomy With an Epidural for Post-Operative Analgesia
Brief Title: IV vs Epidural Opioids + Epidural Local Anesthetic for Laparotomy Analgesia
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Melinda Seering, Clinical Associate Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 202402557
Record Dates: First submitted 2024-07-24; First posted 2024-08-19 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Laparotomy
Keywords: Epidural; PCEA; PCA; Hydromorphone; bupivacaine; analgesia; laparotomy
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient and bedside observer will be blinded to which group the patient is in
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Hydromorphone administered intravenous PCA combined with a continuous bupivacaine epidural infusion
  Interventions: Drug: Intravenous administered opioid
- Treatment (Active Comparator): Hydromorphone combined with bupivacaine in the epidural and administered as a continuous infusion with a PCEA bolus as necessary
  Interventions: Drug: Epidural administered opioid

INTERVENTIONS:
Drug: Intravenous administered opioid — Hydromorphone will be received intravenously using a patient controlled administration pump, as well as patient will have a continuous bupivacaine epidural infusion
  Other Names: hydromorphone IV
  Arms: Control
Drug: Epidural administered opioid — Hydromorphone will be added to the bupivacaine in the epidural and will have a continuous infusion along with the ability for the patient to receive epidural boluses of the medications by a patient controlled epidural administration pump
  Other Names: Hydromorphone epidural
  Arms: Treatment

SUMMARY:
The purpose of this research study is to determine if the two common ways of administering additional opioids (morphine like substance, narcotic) with an epidural, either mixed in the epidural solution or given separately through the intravenous, are equally effective in controlling post-operative pain

DETAILED DESCRIPTION:
Open label, observer and patient blinded randomized control study of patients age 18 to 85 who are booked to have an open upper abdominal surgical incision where an epidural would normally be offered and expected to be used for an average of 4 to 5 days.

Study will be done at University of Iowa Hospitals and Clinics main operating room and post-operative surgical wards.

Eligible patients who choose to consent to participate in the study will be randomized to either have the opioid administered intravenously using patient controlled administration (PCA) device along with a local anesthetic only continuous epidural infusion ,the control group, or to the treatment group of the opioid combined with the local anesthetic in the epidural with a continuous infusion combined with patient controlled epidural administered (PCEA) bolus. The epidural pump along with the PCA machine will be placed in such away that they can be obscured by a removable cover. The patient will be seen daily to obtain pain and satisfaction scores using the Quality of Recovery (QoR) 15. Secondary data will also be collected including presence of side effects, ability to mobilize, signs of return of bowel function, need for supplemental oxygen and total amount of opioid required. Patients will be assigned a study number, which all data will be kept under.

ELIGIBILITY:
Inclusion Criteria:

1. Age including and between 18 to 85 years old
2. Planned open abdominal procedure with an incision that is or includes above the umbilicus, where epidural would normally be offered and epidural would be maintained for an average of 4 to 5 days
3. Patient has consented for an epidural
4. Patient is able to converse in English
5. Patient is able to use a patient controlled pump

Exclusion Criteria:

1. Has a known contraindication for an epidural
2. Known mental or cognitive disability
3. History of chronic opioid use or substance abuse disorder
4. Pre-operative use of opioids
5. History of chronic pain
6. Routine use of marijuana
7. Incarcerated
8. Unable to converse in English
9. Planned to remain intubated post-operatively
10. Need for post-operative use of anticoagulant regiment that would be contraindicated with an indwelling epidural catheter
11. End stage renal disease or dialysis
12. Hepatic disease that affects metabolism of drugs
13. Known contraindication to any of the study drugs
14. Known pregnancy or positive pre-operative pregnancy test
15. Known neurological condition that may affect motor or sensory systems

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
With a local anesthetic epidural, is the epidural administration of opioids similar to opioids administered by intravenous | Once daily until one day after the epidural in discontinued which would mean a maximum of 8 days post-operatively
  Quality of Recovery (QoR) 15 score from 0-150 with the higher the score the better

SECONDARY OUTCOMES:
With a local anesthetic epidural, are there any differences in the incidence of opioid side effects between intravenous and epidural administered opioids | Assessed daily until the epidural is removed, which is maximum of 7 days post-operatively
  will assess patient for symptoms suggestive of opioid side effects and look in the patient's chart to see if they require any medication treatments that could be linked to opioid side effects
Does the route of epidural opioid administration, intravenous vs epidural, affect the return of bowel function | daily assessment until epidural removed, which is a maximum of 7 days post-operatively
  Will assess patient and chart looking for signs of bowel function return and look how patient is able to progress with diet (time in days until signs of bowel function return)
Does the route of epidural opioid administration, intravenous vs epidural, impact patient ability to be discharged | Will follow until patient discharged or maximum 10 days post-operatively
  Will look in chart to see when surgery documents that they feel patient has recovered enough to be discharged home (time in days until dischargeable)

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Seering, MD, Principal Investigator — Univeristy of Iowa
Locations (1):
- University of Iowa Health Care, Iowa City, Iowa, United States